CLINICAL TRIAL: NCT02924194
Title: Deep Brain Stimulation (DBS) of the Nucleus Basalis of Meynert (nbM) to Treat Parkinson's Patients With Mild Cognitive Impairment, Amnestic Subtype
Brief Title: Deep Brain Stimulation of the nbM to Treat Mild Cognitive Impairment in Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was halted prematurely due to lack of interested participants.
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Barrow Neurological Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PHX-16-0141-30-06
Record Dates: First submitted 2016-09-30; First posted 2016-10-05 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Parkinson's Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nbM stimulation ON for 3 months (GPi also on) (Experimental): Subjects will undergo activation of GPi and nbM electrodes The GPi's will be stimulated to achieve improvement in motor function. There is a double blind evaluation of DBS-nbM stimulation. Subjects will be those with nbM stimulation ON for a period of 3 months (GPi also on). No usual treatment is withheld. PD drug doses will be stable unless disabling dyskinesias warrants a reduction of medication. After initial 3 months period of stimulation subject will undergo a repeat of neuropsychological testing and Motor Unified Parkinson's Disease Rating Scale (UPDRS) rating prior to switching group assignment (cross-over). There will be a 2 day wash-out period of nbM stimulation for all subjects (both the On and Off groups) in order to minimize subject bias. Then, the subjects will undergo additional brief neuropsychological testing to asses for carry over effects. The subjects will then be switched to the alternate nbM stimulation group (cross-over) from their previous 3 month period.
  Interventions: Device: stimulation ON
- nbM stimulation OFF for 3 months (GPi is on) (Experimental): Subjects will undergo activation of GPi and nbM electrodes The GPi's will be stimulated to achieve improvement in motor function. There is a double blind evaluation of DBS-nbM stimulation. Subjects will be those with nbM stimulation OFF for a period of 3 months (GPi is on). No usual treatment is withheld. PD drug doses will be stable during blinded parts of the assessment unless disabling dyskinesias warrants a reduction of medication. After initial 3 months period of stimulation subject will undergo a repeat of neuropsychological testing and Motor UPDRS rating prior to switching group assignment (cross-over). There will be a 2 day wash-out period of nbM stimulation for all subjects (both the On and Off groups) in order to minimize subject bias. Then, the subjects will undergo additional brief neuropsychological testing to asses for carry over effects. The subjects will then be switched to the alternate nbM stimulation group (cross-over) from their previous 3 month period.
  Interventions: Device: stimulation OFF

INTERVENTIONS:
Device: stimulation ON — The system used in the study includes the Model 37601 Activa PC stimulator, Model 3387 Lead and Model 37085 Extension, all manufactured and commercially available by Medtronic, Inc. Collectively, these devices will be referred to as "the DBS System". The DBS System is commercially available in the United States and was approved by FDA on July 31, 1997 under PMA P960009. It is indicated for deep brain stimulation for the treatment of symptoms of Parkinson's disease and essential tremor.
  Arms: nbM stimulation ON for 3 months (GPi also on)
Device: stimulation OFF — The system used in the study includes the Model 37601 Activa PC stimulator, Model 3387 Lead and Model 37085 Extension, all manufactured and commercially available by Medtronic, Inc. Collectively, these devices will be referred to as "the DBS System". The DBS System is commercially available in the United States and was approved by FDA on July 31, 1997 under PMA P960009. It is indicated for deep brain stimulation for the treatment of symptoms of Parkinson's disease and essential tremor.
  Arms: nbM stimulation OFF for 3 months (GPi is on)

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of deep brain stimulation of the nucleus basalis of Meynert (also called the "nbM") at improving memory in Parkinson's disease patients with mild cognitive impairments and memory difficulties. Patients with Parkinson's disease (PD) that are eligible for Deep Brain Stimulation (DBS) therapy for improvement of their motor symptoms and with evidence of mild cognitive impairments and memory difficulties will be enrolled.

DETAILED DESCRIPTION:
This is a prospective, double-blind (patient and neuropsychologist), randomized, cross-over study to evaluate the safety of deep brain stimulation of the nucleus basalis of Meynert (nbM) in Parkinson's disease (PD) patients with mild cognitive impairment (PD-MCI) who are undergoing globus pallidus internus (GPi) stimulation for their motor symptoms. Six patients with PD who are eligible for GPi DBS for improvement of their motor symptoms and who have a clinical diagnosis of PD-MCI (amnestic, single or multiple domain) per Movement Disorder Society (MDS) criteria will be enrolled and implanted with bilateral electrodes in in the nbM in addition to the globus pallidus internus (GPi). Conventional stereotactic implantation of the electrodes will be guided by intraoperative computerized tomography (CT) and magnetic resonance tomography (MRT).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed by the subject.
* Parkinson's disease per UK Parkinson's Disease Society Brain Bank (Queens Square) criteria
* Diagnosis of PD-MCI, amnestic subtype per MDS criteria (Level II assessment)
* DBS candidate for GPi targeting per the consensus committee
* 50 - 75 years of age
* Primary English speaking
* Minimum of 10 years of education
* Motorically and cognitively capable of completing evaluations and consent
* Medically cleared for surgery and anesthesia
* Subject must be on stable doses of any medication used to treat PD or cognition for 3 months prior to study entry
* Female subjects with child-bearing potential have a negative serum pregnancy test prior to DBS surgery -

Exclusion Criteria:

* Dementia per DSM-V criteria
* Condition precluding MRI
* History of supraspinal CNS disease other than PD
* Medical condition or required medication compromising cognition
* Alcohol use of more than 4 drinks per day
* Currently uncontrolled moderate-severe depression (BDI>20)
* History of suicide attempt in the year preceding study screening
* History of schizophrenia, delusions, or currently uncontrolled visual hallucinations
* Use of cholinesterase inhibitor
* Subjects who require rTMS, ECT, diathermy, or repeat MRI procedures to treat a medical condition.
* Subjects with a history of seizure disorder
* Subjects who have made a suicide attempt within the prior year,
* Subjects with any medical contraindications to undergoing DBS surgery (eg, infection, coagulopathy, or significant cardiac or other medical risk factors for surgery)
* Subjects with an implanted stimulator such as a cardiac pacemaker, defibrillator, neurostimulator and cochlear implant
* Subjects who are pregnant or nursing.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-09; Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Evaluate safety of DBS-nbM | Month 36
  Evaluate safety through collection of adverse events at weeks 4, 16, 28, 52 and months 24 and 36.

SECONDARY OUTCOMES:
Stability or improvement of cognitive symptoms | Month 36
  Administration of Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) administered at Week 52 and Months 24 and 36. A clinically meaningful change is indicated by a 4 point change in ADAS-Cog.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco A Ponce, MD, Principal Investigator — Barrow Brain and Spine
Locations (1):
- St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No